CLINICAL TRIAL: NCT03861533
Title: Guidelines Oriented Approach to Lipid Lowering Quality Enhancement Research Initiative (GOAL QuERI) International
Brief Title: GOAL International QuERI - Protocol CHRC 2019 GOAL INTERNATIONAL
Acronym: GOAL QuERI
Status: Completed | Type: Observational
Sponsor: Dr. Anatoly Langer (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Dr. Anatoly Langer, MD, M.Sc., FRCP (C), FACC, Canadian Heart Research Centre
Organization: Canadian Heart Research Centre (Other)
Other Study IDs: CHRC2019-GOAL INT
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Surveys and Questionnaires; Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey — Cross-Reference
  Other Names: cross-sectional study without specific intervention

SUMMARY:
This Quality Enhancement Research Initiative (QuERI) is a knowledge translation medical practice activity based on decision making support through feedback to physicians on their management of dyslipidemia in order to achieve guidelines recommended LDL-C levels in high risk patients. Physician interaction has three distinct components:

1. Capture of data as reported by participating physician;
2. Highlight (by providing feedback) where management may be optimized based on guidelines or recommendations;
3. Identify challenges faced by physicians resulting in the care gap..

DETAILED DESCRIPTION:
The GOAL QuERI International will engage approximately 115 health care practitioners (HCP) who will enroll up to 2500 patients with management observations based on four visits by the patients in an outpatient setting. The timing of the visits will be baseline, 6±2 months, 12±2 months, and 18±2 months during which patient management by their physician will be captured using the electronic data capture form (DCF). The DCF will be created and managed by the CHRC.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years old
2. High risk for cardiovascular morbidity and mortality such as prior history of clinical cardiovascular disease and/or history of familial hypercholesterolemia
3. LDL-C within the past 6 months above recommended level despite maximal tolerated statin therapy ± ezetimibe for the past 3 months.

Exclusion Criteria:

1. Current treatment with PCSK9 inhibitor
2. Current participation in investigational study
3. Prior participation in the GOAL program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GOAL International enrolling approximately 2500 patients with clinical vascular disease or familial hypercholesterolemia (FH) and LDL-C > 2.0 mmol/L (77 mg/dl) despite maximally tolerated statin therapy. As part of an interactive knowledge translation component, physicians are asked to indicate their next steps in lowering of LDL-C and are then asked whether they will be following the guidelines and if not why not.
Sampling Method: Non-Probability Sample
Enrollment: 2422 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving country specific guideline-recommended LDL-C levels after 18 month final visit or last available observation during follow up visits. | LDL-C target after 18 month final visit
  the outcome variable, LDL-C, will be presented with mean and standard deviation

SECONDARY OUTCOMES:
1. Relative and absolute reduction of LDL-C with lipid lowering medications added during the observation period. | The timing of the visits will be baseline, 6±2 months, 12±2 months, and 18±2 months during which patient management by their physician will be captured using the electronic data capture
  the outcome variable, LDL-C, will be presented with mean and standard deviation
Proportion of patients not achieving recommended LDL-C level based on high risk inclusion sub-group (e.g. FH), co-morbid conditions (diabetes mellitus), baseline treatment or baseline lipid profile. | The timing of the visits will be baseline, 6±2 months, 12±2 months, and 18±2 months during which patient management by their physician will be captured using the electronic data capture
  the outcome variable, LDL-C, will be presented with mean and standard deviation
Proportion of patients not achieving recommended LDL-C level at each of the follow up visits according to physician responses as to why country specific recommendation for LDL-C lowering opportunities was not followed. | The timing of the visits will be baseline, 6±2 months, 12±2 months, and 18±2 months during which patient management by their physician will be captured using the electronic data capture
  the outcome variable, LDL-C, will be presented with mean and standard deviation
Proportion of patients achieving LDL-C and non-HDL level across participating countries. | The timing of the visits will be baseline, 6±2 months, 12±2 months, and 18±2 months during which patient management by their physician will be captured using the electronic data capture
  the outcome variable, LDL-C, will be presented with mean and standard deviation

CONTACTS AND LOCATIONS:
Overall Officials: Anatoly Langer, MD, M.Sc, FRCP(C,) FACC, Study Chair — Canadian Heart Rersearch Centre
Locations (4):
- Sabah Hosptial, Kuwait City, Kuwait
- Centro de Estudios Clínicos de Querétaro (CECLIQ), Querétaro City, Querétaro, Mexico
- King Fahd Military Medical Complex, Dhahran, Saudi Arabia
- Cleveland Clinic, Abu Dhabi, United Arab Emirates